CLINICAL TRIAL: NCT03987113
Title: Impact of Cold Ischemia on Pulmonary Endothelial Dysfunction in Ex-vivo Pulmonary Reconditioning
Acronym: Endoth-Exvivo
Status: Completed | Type: Observational
Sponsor: Hopital Foch (Other)
Collaborators: Institut National de la Santé Et de la Recherche Médicale Rouen U1096 (Unknown)
Responsible Party: Sponsor
Other Study IDs: 2017022F
Record Dates: First submitted 2019-06-12; First posted 2019-06-14 (Actual); Last update posted 2020-07-14 (Actual); Status verified 2019-07

CONDITIONS: Lung Transplant

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Plasma concentration analysis during and after ex-vivo pulmonary reconditioning — The pulmonary endothelial dysfunction will be evaluated with plasma concentration of heparan sulphate, syndecan-1, endothelin-1 and i-NOS.

SUMMARY:
The study population will be patients with planned double-lung transplant, with preoperative ex-vivo reconditioning procedure.

The ex-vivo procedure will be performed for lungs considered as limit to be directly implanted according to the national classification or in case of Maastrich 3 decision. They required a rehabilitation procedure like ex-vivo to determine their quality. Once the procedure initiated, the unused remaining liquid will be retrieved for the first gasometry usually performed. This will be the time T1 of sampling.

The unused remaining liquid will be retrieved for the gasometry of end of procedure usually performed, before the graft cooling. This will be the time T2.

The purge liquid of first lung at the declamping of the pulmonary artery will be retrieved at the time of unclamping (time T3 of sampling).

The purge liquid of the second lung at the declamping of the pulmonary artery will be retrieved with the same procedure (time T4 of sampling).

The samples will be analysed with ELISA technique. The endothelial dysfunction will be evaluated with plasma concentration of heparan sulphate, syndecan-1, endothelin-1 and i-NOS.

ELIGIBILITY:
Selection Criteria:

* patient aged > 18 years old
* patient with healthcare insurance
* non-opposition of the patient
* patient with usual criteria for lung transplant and planned lung transplant after meeting of staff transplant

Non Selection Criteria:

* participation refusal
* patient under tutorship or guardianship
* protected adult

Inclusion Criteria:

* selected patient with Biomedecine Agency agreement for graft allocation off tour

Exclusion Criteria:

* selected patient with Biomedicine Agency agreement for standard allocation graft

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient who requires a lung transplant, with ex-vivo reconditioning procedure. The objective is to create a plasma bank for all these patients with post analysis of sample.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2018-11-15 (Actual); Primary Completion 2019-10-30 (Actual); Study Completion 2019-10-30 (Actual)

PRIMARY OUTCOMES:
Correlation between time of cold ischemia and endothelial dysfunction | 24 hours
  Plasma concentration in heparin sulphate, syndecan-1, endothelin-1 and i-NOS

SECONDARY OUTCOMES:
Correlation between time of cold ischemia and systemic inflammation | 24 hours
  Plasma concentration in IL-1β, IL-8, IL-10 and TNF-α

CONTACTS AND LOCATIONS:
Overall Officials: Morgan LE GUEN, Principal Investigator — Anaesthesia department
Locations (1):
- Hôpital Foch, Suresnes, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Selim J, Wolf J, Soulie M, Sage E, Glorion M, Fessler J, Mulder P, Vasse M, Bellien J, Djerada Z, Richard V, Guen ML. Post-Ex Vivo Lung Perfusion Hypothermic Storage Limits Inflammation and Endothelial Dysfunction. J Cardiothorac Vasc Anesth. 2025 Oct;39(10):2748-2759. doi: 10.1053/j.jvca.2025.07.007. Epub 2025 Jul 8. PMID 40738815